CLINICAL TRIAL: NCT05357079
Title: The Impact of Topical Tranexamic Acid on Pre- and Post-operative Hemoglobin / Hematocrit in Isolated Operative Posterior Wall Acetabular Fractures: a Prospective, Randomized, Double-blinded, Multicenter Study
Brief Title: Impact of Topical Tranexamic Acid on Pre- and Post-operative Hemoglobin/Hematocrit
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Foundation for Orthopedic Trauma (Unknown)
Responsible Party: Principal Investigator, Michael Archdeacon, Professor & Chair, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 2016-2519
Record Dates: First submitted 2021-07-20; First posted 2022-05-02 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-12

CONDITIONS: Fracture of Posterior Wall of Acetabulum
MeSH Terms: interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: A. Specific aims
  a. To conduct a multi-center study to prospectively evaluate the use of topical tranexamic acid (TXA - Cyklokapron; Pfizer, New York, NY) on pre-operative and post-operative hemoglobin (Hb)/hematocrit (Hct) in patients undergoing operative repair of isolated posterior wall (PW) acetabular fractures.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical TXA Treatment (Experimental): 2 gm TXA/100 ml of normal saline
  Interventions: Drug: Tranexamic Acid
- No Topical Treatment (Placebo Comparator): Normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic Acid — Topical application
  Other Names: Cyklokapron, Pfizer
  Arms: Topical TXA Treatment
Drug: Normal saline — Topical application
  Arms: No Topical Treatment

SUMMARY:
This multi-center, prospective study will evaluate the use of topical tranexamic acid (TXA - Cyklokapron; Pfizer, New York, NY) on pre-operative and post-operative hemoglobin (Hb)/hematocrit (Hct) in patients undergoing operative repair of isolated posterior wall (PW) acetabular fractures.

DETAILED DESCRIPTION:
In this prospective, randomized, double-blinded, multi-center study comparing topical TXA with placebo, investigators will determine whether topical TXA utilization in isolated PW acetabular surgery has beneficial or detrimental effects.

In order to evaluate the delta between pre-operative and post-operative hemoglobin (blood loss parameters) in patients with isolated PW acetabular fractures that were treated with topical TXA or a placebo, investigators will prospectively enroll all eligible patients with the diagnosis of a closed, isolated, PW acetabular fracture that requires surgical fixation. Isolated PW fractures have been chosen to reduce confounding variables, particularly those associated with more complex fracture patterns including longer surgery duration and blood loss.

Each subject will have a pre-operative Hb and Hct drawn on the morning of surgery to establish a baseline level. Prior to surgery, subjects will be computer-randomized by pharmacy to one of two groups: a topical TXA group and a control group. The topical TXA group will be treated with 2 gm/100 ml of normal saline, while the control group will be treated with a placebo (normal saline) in a similar fashion to the TXA experimental group.

The surgeon and the operative team will be blinded as to whether the patient receives TXA or placebo.

Intraoperative transfusion requirements and estimated blood loss (EBL) will be recorded for every patient.

Hemoglobin and hematocrit values will be obtained on postoperative day one and two with routine morning blood draws (typically 5 am-9 am). Post-operative transfusion requirements prior to discharge will be recorded. All patients will have standard low molecular weight heparin DVT prophylaxis for four weeks post-operatively.

Prospectively demographic data will be collected. Injury and treatment data collected will include date of injury, mechanism of injury, laterality of injury, medical co-morbidities, associated injuries, date of surgery, operative time, estimated operative blood loss (EBL) from both anesthesia and operative surgeon, calculated operative blood loss, as well as hemoglobin/hematocrit as described, and blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an isolated, closed, posterior wall acetabular fracture managed surgically within 7 days of injury. Upper extremity fractures that are non-operative and have no impact on weight-bearing status will be included.
2. Patients must be skeletally mature.

Exclusion Criteria:

1. Patients are not skeletally mature.
2. Patients with any concomitant lower extremity, pelvis, or spine injuries.
3. Patient admitted as a polytrauma patient to the trauma service due to injury to an internal organ (head, chest, or abdomen).
4. Patient has an unidentified source of hemorrhage other than acetabular fracture.
5. Patient requires surgery for treatment of concomitant injuries.
6. Patient requires multiple surgeries.
7. Patient has pre-existing thrombus prior to surgery.
8. Patient with a history of prior pulmonary embolus or other thromboembolic disease.
9. Patient with a known bleeding disorder.
10. Patient with a history of renal insufficiency.
11. Patient who is unable to give consent or is unconscious.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (Hb) | Postoperative Day 2
  Hemoglobin (Hb) results
Hematocrit (Hct) | Postoperative Day 2
  Hematocrit (Hct) results

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati College of Medicine, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magnussen RA, Tressler MA, Obremskey WT, Kregor PJ. Predicting blood loss in isolated pelvic and acetabular high-energy trauma. J Orthop Trauma. 2007 Oct;21(9):603-7. doi: 10.1097/BOT.0b013e3181599c27. PMID 17921834
- [Background] Lemaire R. Strategies for blood management in orthopaedic and trauma surgery. J Bone Joint Surg Br. 2008 Sep;90(9):1128-36. doi: 10.1302/0301-620X.90B9.21115. PMID 18757950
- [Background] Hiippala ST, Strid LJ, Wennerstrand MI, Arvela JV, Niemela HM, Mantyla SK, Kuisma RP, Ylinen JE. Tranexamic acid radically decreases blood loss and transfusions associated with total knee arthroplasty. Anesth Analg. 1997 Apr;84(4):839-44. doi: 10.1097/00000539-199704000-00026. PMID 9085968
- [Background] Yamasaki S, Masuhara K, Fuji T. Tranexamic acid reduces postoperative blood loss in cementless total hip arthroplasty. J Bone Joint Surg Am. 2005 Apr;87(4):766-70. doi: 10.2106/JBJS.D.02046. PMID 15805205
- [Background] Ralley FE, Berta D, Binns V, Howard J, Naudie DD. One intraoperative dose of tranexamic Acid for patients having primary hip or knee arthroplasty. Clin Orthop Relat Res. 2010 Jul;468(7):1905-11. doi: 10.1007/s11999-009-1217-8. Epub 2010 Jan 9. PMID 20063079
- [Background] Phillips SJ, Chavan R, Porter ML, Kay PR, Hodgkinson JP, Purbach B, Reddick AH, Frayne JM. Does salvage and tranexamic acid reduce the need for blood transfusion in revision hip surgery? J Bone Joint Surg Br. 2006 Sep;88(9):1141-2. doi: 10.1302/0301-620X.88B9.17605. PMID 16943461
- [Background] Johansson T, Pettersson LG, Lisander B. Tranexamic acid in total hip arthroplasty saves blood and money: a randomized, double-blind study in 100 patients. Acta Orthop. 2005 Jun;76(3):314-9. PMID 16156456
- [Background] Kelley TC, Tucker KK, Adams MJ, Dalury DF. Use of tranexamic acid results in decreased blood loss and decreased transfusions in patients undergoing staged bilateral total knee arthroplasty. Transfusion. 2014 Jan;54(1):26-30. doi: 10.1111/trf.12167. Epub 2013 Mar 22. PMID 23521109
- [Background] Piggott RP, Leonard M. Is there a role for antifibrinolytics in pelvic and acetabular fracture surgery? Ir J Med Sci. 2016 Feb;185(1):29-34. doi: 10.1007/s11845-015-1375-5. Epub 2015 Nov 11. PMID 26560109
- [Background] Ho KM, Ismail H. Use of intravenous tranexamic acid to reduce allogeneic blood transfusion in total hip and knee arthroplasty: a meta-analysis. Anaesth Intensive Care. 2003 Oct;31(5):529-37. doi: 10.1177/0310057X0303100507. PMID 14601276
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Zufferey PJ, Miquet M, Quenet S, Martin P, Adam P, Albaladejo P, Mismetti P, Molliex S; tranexamic acid in hip-fracture surgery (THIF) study. Tranexamic acid in hip fracture surgery: a randomized controlled trial. Br J Anaesth. 2010 Jan;104(1):23-30. doi: 10.1093/bja/aep314. PMID 19926634
- [Background] Wei W, Wei B. Comparison of topical and intravenous tranexamic acid on blood loss and transfusion rates in total hip arthroplasty. J Arthroplasty. 2014 Nov;29(11):2113-6. doi: 10.1016/j.arth.2014.07.019. Epub 2014 Jul 30. PMID 25155138
- [Background] Patel JN, Spanyer JM, Smith LS, Huang J, Yakkanti MR, Malkani AL. Comparison of intravenous versus topical tranexamic acid in total knee arthroplasty: a prospective randomized study. J Arthroplasty. 2014 Aug;29(8):1528-31. doi: 10.1016/j.arth.2014.03.011. Epub 2014 Mar 21. PMID 24768543
- [Background] Dailey SK, Archdeacon MT. Open reduction and internal fixation of acetabulum fractures: does timing of surgery affect blood loss and OR time? J Orthop Trauma. 2014 Sep;28(9):497-501. doi: 10.1097/BOT.0000000000000153. PMID 24824098
- [Background] Furey AJ, Karp J, O'Toole RV. Does early fixation of posterior wall acetabular fractures lead to increased blood loss? J Orthop Trauma. 2013 Jan;27(1):2-5. doi: 10.1097/BOT.0b013e31824d96de. PMID 22495528
- [Background] Lisander B, Ivarsson I, Jacobsson SA. Intraoperative autotransfusion is associated with modest reduction of allogeneic transfusion in prosthetic hip surgery. Acta Anaesthesiol Scand. 1998 Jul;42(6):707-12. doi: 10.1111/j.1399-6576.1998.tb05305.x. PMID 9689278
- [Background] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146
- [Background] Tornetta P 3rd. Non-operative management of acetabular fractures. The use of dynamic stress views. J Bone Joint Surg Br. 1999 Jan;81(1):67-70. doi: 10.1302/0301-620x.81b1.8805. PMID 10068006